CLINICAL TRIAL: NCT05303038
Title: A Phase II Clinical Study of Cryoablation Combined With Tirelizumab and Bevacizumab in Liver Metastatic Triple Negative Breast Cancer Patients Failed by Multiline Therapy
Brief Title: Cryoablation Combined With Tirelizumab and Bevacizumab in Liver Metastatic TNBC Patients Failed by Multiline Therapy
Acronym: Castle06(BC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Castle06(BC)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer in the Liver
Keywords: Triple Negative Breast Cancer; Cryoablation; Tirelizumab; Bevacizumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cryoablation combined with tirelizumab + Bevacizumab (Experimental)
  Interventions: Combination Product: Cryoablation Combined with Tirelizumab and Bevacizumab

INTERVENTIONS:
Combination Product: Cryoablation Combined with Tirelizumab and Bevacizumab — Cryoablation of 1-2 typical metastatic lesions will be performed on D1 under general anesthesia and ultrasound guidance for two cycles.
  200mg Tirelizumab ( IV Q3W) + Bevacizumab 7.5mg/kg ( IV Q3W) will be administered at D14 after cryoablation.

SUMMARY:
This is a Phase II, open-label study evaluating the efficacy and safety of Cryoablation combined with Tirelizumab and Bevacizumab in liver metastatic triple-negative breast cancer patients failed by multiline therapy.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center phase II clinical trial in liver metastatic triple-negative breast cancer patients failed by multiline therapy.

All subjects will receive cryoablation combined with tirelizumab + bevacizumab:

1. Cryoablation of liver metastases: Cryoablation of 1-2 typical metastatic lesions will be performed on D1 under general anesthesia and ultrasound guidance for two cycles. If the patient has no measurable lesions outside the liver, the measurable lesions should be retained after partial ablation of the liver lesions.
2. PD-1 antibody + anti vascular therapy: patients will receive 200mg Tirelizumab ( IV Q3W) + Bevacizumab 7.5mg/kg ( IV Q3W) at D14 after cryoablation until there is disease progression, intolerable toxic reaction, subject withdraws informed consent or the study ends (whichever comes first).
3. Puncture biopsy of liver metastases will completed 1-3 days before cryoablation, 1-3 days before the first treatment with tirelizumab + bevacizumab, 2 cycles after treatment with tirelizumab + bevacizumab and after disease progression, and blood samples (about 10ml) were collected for mutation load detection and immune function evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or Imageologically confirmed liver metastatic tnbc patients;
* Histologically confirmed diagnosis of TNBC characterized by estrogen receptor negative (ER-), progesterone receptor negative (PR-) and human epidermal growth factor-2 receptor negative (HER2-);
* ≥ 2 prior lines systemic therapy;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1);
* The patients show no signs of bile duct obstruction, and the bilirubin is below the upper limit of 1.5x normal value (ULN);
* Age ≥ 18 years on the day of signing the ICF (or the legal age of consent in the jurisdiction in which the study is taking place);
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* The functions of the patient's organs and blood system meet the requirements;
* Blood system function: absolute neutrophil count (ANC) ≥ 1.5 x 109 / L, platelet count ≥ 100 x 109 / L
* Renal function: estimated glomerular filtration rate or creatinine clearance > 50 ml / min / 1.73 M2
* Liver function: total bilirubin ≤ 1.5 x ULN, AST and alt ≤ 5 x ULN
* Estimated survival time ≥12 weeks.

Exclusion Criteria:

* The patient is currently receiving or has received irradiation or local treatment for the target lesion in the past 3 weeks.
* The patient had previously received cryoablation.
* The patient received major surgery within 14 days before enrolling in the study.
* Palliative radiotherapy must be completed at least 2 weeks before enrolling in the study, and there is no plan for additional radiotherapy for the same lesion; ·Patients whose AE caused by radiotherapy did not recover to ≤ CTCAE 1 degree
* The patient had metastatic brain lesions, including asymptomatic and well controlled lesions.
* Complicated with infection and requiring intravenous antibiotic treatment.
* The patient has any clinically significant disease or history that the investigator believes may endanger the safety of the patient or the reliability of the study results.
* The patient has a history of any other malignancy unless the remission period exceeds 1 year. (do not exclude skin cancer, cervical cancer in situ, superficial bladder cancer, and breast cancer in radical treatment).
* Female patients are pregnant or breastfeeding.
* The patient received any trial drug within 14 days before receiving the first study drug.
* The patient had undiminished or unstable severe toxicity (≥ CTCAE 4.0 grade 2) after previous use of another trial drug and / or previous cancer treatment, except anemia, weakness and hair loss.
* Patients are allergic to the test drug or any of its excipients.
* Patients are known to be HIV positive, have HCB, or have HBV infection and HBV DNA exceeds 2000 IU / ml.
* The patient has a known history of drug addiction in the past 1 year, because this situation may lead to a high risk of non-compliance of the trial drug.
* The patient has known active or suspected autoimmune disease. Subjects who are in a stable state and do not need systemic immunosuppressive therapy are allowed to be enrolled.
* Subjects requiring systemic treatment with corticosteroids (> 10mg / day prednisone efficacy dose) or other immunosuppressants within 14 days before the administration of the study drug were allowed to inhale or locally use steroids and adrenal hormone replacement with a dose > 10mg / day prednisone efficacy dose in the absence of active autoimmune diseases.
* The patient had a baseline corrected QT interval QTc > 450 ms, or the patient had known QT prolongation syndrome, torsade de pointe ventricular tachycardia, symptomatic ventricular tachycardia, unstable heart syndrome within 3 months before the screening visit, > grade 2 New York Heart Association heart failure, > grade 2 Canadian Cardiovascular Association angina pectoris.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 12 months
  The number of people with tumor responses according to RECIST (V1.1): the proportion of participants who achieves a best overall response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 12 months
  The time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Disease Control Rate (DCR) | Up to 12 months
  The proportion of participants who achieves a best overall response of CR, PR or stable disease(SD).
Progression-free Survival (PFS) | Up to 12 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.
One-year overall survival (OS) rate | Up to 12 months
  OS defined as the time from the date of randomization to the date of death due to any reason. One-year survival rate (percentage of subjects alive at 1 year) was estimated from OS data.
Frequencies of Biomarkers | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Shangshai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided